CLINICAL TRIAL: NCT05403424
Title: Investigation of Biomechanical and Viscoelastic Properties of Thoracolumbar Fascia in Pregnant Women With Pelvic Girdle Pain
Brief Title: Biomechanical and Viscoelastic Properties of Thoracolumbar Fascia in Pregnancy Pelvic Girdle Pain
Status: Recruiting | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 33 09/03/2022
Record Dates: First submitted 2022-04-15; First posted 2022-06-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pregnant Women; Pelvic Girdle Pain
Keywords: pregnant women; pelvic girdle pain; thoracolumbar fascia; stiffness; creep
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Pregnant women with pelvic girdle pain: This group will consist of pregnant women diagnosed with pelvic girdle pain.
  Interventions: Other: Evaluation of pain; Diagnostic Test: Application of pelvic girdle diagnostic tests; Other: Evaluation of biomechanics and viscoelastic properties of thoracolumbar fascia; Other: Evaluation of activity limitation
- Group 2: Pregnant women without pelvic girdle pain: This group will consist of pregnant women who do not have pelvic girdle pain.
  Interventions: Other: Evaluation of pain; Diagnostic Test: Application of pelvic girdle diagnostic tests; Other: Evaluation of biomechanics and viscoelastic properties of thoracolumbar fascia; Other: Evaluation of activity limitation
- Group 3: Non-pregnant women: This group will consist of non-pregnant women.
  Interventions: Other: Evaluation of biomechanics and viscoelastic properties of thoracolumbar fascia

INTERVENTIONS:
Other: Evaluation of pain — The severity of pelvic girdle pain will be evaluated with the Visual Analog Scale (VAS).
  Groups: Group 1: Pregnant women with pelvic girdle pain; Group 2: Pregnant women without pelvic girdle pain
Diagnostic Test: Application of pelvic girdle diagnostic tests — Pelvic girdle pain diagnostic tests will be applied.
  Groups: Group 1: Pregnant women with pelvic girdle pain; Group 2: Pregnant women without pelvic girdle pain
Other: Evaluation of biomechanics and viscoelastic properties of thoracolumbar fascia — The biomechanical and viscoelastic properties of the thoracolumbar fascia will be measured in the prone position and measurements will be taken from three different points
Other: Evaluation of activity limitation — Pelvic Girdle Questionnaire will be filled
  Groups: Group 1: Pregnant women with pelvic girdle pain; Group 2: Pregnant women without pelvic girdle pain

SUMMARY:
It has not been objectively clarified how the thoracolumbar fascia (TLF) changes the biomechanical adaptations that occur in the lumbopelvic region during pregnancy and whether it is associated with pelvic girdle pain (PGP). Therefore, the aim of this study is to determine the biomechanical and viscoelastic properties of TLF, which adapts to the changes in the lumbopelvic region in pregnant women with pelvic girdle pain, and to investigate its relationship with PGP.

ELIGIBILITY:
Inclusion Criteria:

* First-time pregnancy
* Pregnant women diagnosed with pelvic girdle pain in 1st and 2nd trimesters
* Pregnant women who do not have pelvic girdle pain in 1st and 2nd trimesters
* Women not being pregnant
* Pre-pregnancy Body-Mass-Index (BMI) < 30 kg/m2

Exclusion Criteria:

* Presence of connective tissue disease
* Deterioration of skin integrity in measurement areas
* Presence of orthopedic, neurological, rheumatic problems that may cause musculoskeletal disorders and deviations from normal biomechanical alignment
* History of spine, pelvis, or lower extremity surgery or fracture in the past 6 months
* Definition of chronic low back-pelvic region pain (lasting for more than 3 months and pain severity >4 according to VAS) before pregnancy
* Identification of metabolic disorders such as Type I, II diabetes, gestational diabetes mellitus (GDM), preeclampsia before and/or during pregnancy)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women Healty Women
Study Population: Pregnant women with and without PGP and non-pregnant women
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of biomechanical properties of thoracolumbar fascia | Measurement the change from baseline stiffness values of Thoracolumbar fascia at 12. week and at 22. week
  Measuring of the stiffness (N/m) of the thoracolumbar fascia (with MyotonPro, Myoton AS, Tallin, Estonia) in the prone position.
Evaluation of biomechanical properties of thoracolumbar fascia | Measurement the change from baseline decrement values of Thoracolumbar fascia at 12. week and at 22. week
  Measuring of the decrement of the thoracolumbar fascia (with MyotonPro, Myoton AS, Tallin, Estonia) in the prone position.
Evaluation of biomechanical properties of thoracolumbar fascia | Measurement the change from baseline tone values of Thoracolumbar fascia at 12. week and at 22. week
  Measuring of the tone (Hz) of the thoracolumbar fascia (with MyotonPro, Myoton AS, Tallin, Estonia) in the prone position.
Evaluation of viscoelastic properties of thoracolumbar fascia | Measurement the change from baseline creep values of Thoracolumbar fascia at 12. week and at 22. week
  Measuring of the creep of the thoracolumbar fascia (with MyotonPro, Myoton AS, Tallin, Estonia) in the prone position.
Evaluation of viscoelastic properties of thoracolumbar fascia | Measurement the change from baseline relaxation time values of Thoracolumbar fascia at 12. week and at 22. week
  Measuring of thethe relaxation time (ms) of the thoracolumbar fascia (with MyotonPro, Myoton AS, Tallin, Estonia) in the prone position.

SECONDARY OUTCOMES:
Determining of painful areas | Baseline
  Marking of body chart
Evaluation of pain | Baseline
  Pain will be evaluated with Visual analog scale (VAS). The VAS is scaled between 0-10 points (0: no pain, 10: most severe pain).
Application of Pelvic Girdle Pain (PGP) diagnostic tests | Baseline
  The PGP diagnostic tests will be applied. The posterior pelvic pain provocation test is a pain provocation test used to determine the presence of sacroiliac dysfunction. No score is defined for tests.
Pelvic Girdle Questionnaire | Baseline
  Activity limitation will be evaluated Pelvic Girdle Questionnaire
Evaluation of Body Weight | Measurement the change from baseline body weight (kg) at 12. and 22. weeks.
  Measuring of the Body Weight
Evaluation of Body Mass Index (BMI) | Measurement the change from baseline BMI values at 12.and 22. weeks
  BMI (kg/m2) will be calculated as person's weight in kilograms divided by the square of height in meters.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Alcaraz-Clariana S, Garcia-Luque L, Garrido-Castro JL, Carmona-Perez C, Rodrigues-de-Souza DP, Fernandez-de-Las-Penas C, Alburquerque-Sendin F. Influence of Spinal Movements Associated with Physical Evaluation on Muscle Mechanical Properties of the Lumbar Paraspinal in Subjects with Acute Low Back Pain. Diagnostics (Basel). 2022 Jan 25;12(2):302. doi: 10.3390/diagnostics12020302. PMID 35204392
- [Result] Aldabe D, Milosavljevic S, Bussey MD. A multivariate model for predicting PPGP considering postural adjustment parameters. Musculoskelet Sci Pract. 2020 Aug;48:102153. doi: 10.1016/j.msksp.2020.102153. Epub 2020 May 5. PMID 32560861
- [Result] Lohr C, Braumann KM, Reer R, Schroeder J, Schmidt T. Reliability of tensiomyography and myotonometry in detecting mechanical and contractile characteristics of the lumbar erector spinae in healthy volunteers. Eur J Appl Physiol. 2018 Jul;118(7):1349-1359. doi: 10.1007/s00421-018-3867-2. Epub 2018 Apr 20. PMID 29679246
- [Result] Wu Z, Wang Y, Ye Z, Guan Y, Ye X, Chen Z, Li C, Chen G, Zhu Y, Du J, Chen G, Liu W, Xu X. Effects of Age and Sex on Properties of Lumbar Erector Spinae in Healthy People: Preliminary Results From a Pilot Study. Front Physiol. 2021 Sep 20;12:718068. doi: 10.3389/fphys.2021.718068. eCollection 2021. PMID 34616306
- [Result] Stuge B, Garratt A, Krogstad Jenssen H, Grotle M. The pelvic girdle questionnaire: a condition-specific instrument for assessing activity limitations and symptoms in people with pelvic girdle pain. Phys Ther. 2011 Jul;91(7):1096-108. doi: 10.2522/ptj.20100357. Epub 2011 May 19. PMID 21596959